CLINICAL TRIAL: NCT05607680
Title: A Randomized, Double-blind, Placebo-controlled Phase III Study Evaluating the Efficacy and Safety of IBI362 in Chinese Participants With Obesity or Overweight (GLORY-1)
Brief Title: A Study of IBI362 in Participants With Obesity or Overweight
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CIBI362B301
Record Dates: First submitted 2022-10-23; First posted 2022-11-07 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Obesity Or Overweight
MeSH Terms: interventions — mazdutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo,SC,once a week for 48 weeks
  Interventions: Drug: Placebo
- IBI362 4 mg (Experimental): 2 mg,SC,once a week for 4 weeks 4 mg,SC,once a week for 44 weeks
  Interventions: Drug: IBI362
- IBI362 6 mg (Experimental): 2 mg,SC,once a week for 4 weeks 4 mg,SC,once a week for 4 weeks 6 mg,SC,once a week for 40 weeks
  Interventions: Drug: IBI362

INTERVENTIONS:
Drug: Placebo — Placebo administered subcutaneously (SC) once a week.
  Arms: Placebo
Drug: IBI362 — IBI362 administered subcutaneously (SC) once a week.
  Arms: IBI362 4 mg; IBI362 6 mg

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled Phase III clinical study evaluating the efficacy and safety of IBI362 in overweight or obese subjects. Subjects will be randomly assigned to IBI362 low-dose, high-dose and placebo groups. The entire trial cycle includes a 2-week screening period, a 48-week double-blind treatment period, and a 12-week drug withdrawal follow-up period after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

• Body mass Index (BMI) ≥28 kilograms per square meter (kg/m²), or ≥24 kg/m² and with at least one of the following comorbidities: prediabetes, hypertension, dyslipidemia, fatty liver, weight bearing joint pain, obesity-related dyspnea or obstructive sleep apnea.

Exclusion Criteria:

* HbA1c ≥ 6. 5% at screening or previous diagnosis of type 1 or type 2 diabetes;
* Weight change > 5.0% after diet and exercise control for at least 12 weeks before screening;
* Have used or are currently using weight loss drugs within 3 months before screening;
* History of pancreatitis;
* Family or personal history of thyroid C-cell carcinoma or multiple endocrine neoplasia (MEN) 2A or 2B；
* History of moderate to severe depression or severe mental illness;
* Any lifetime history of a suicide attempt

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline, Week 32
Percentage of Participants who Achieve ≥5% Body Weight Reduction | Week 32

SECONDARY OUTCOMES:
Percentage of Participants who Achieve ≥10%Body Weight Reduction | Week 32,Week 48
Percentage of Participants who Achieve ≥15% Body Weight Reduction | Week 32,Week 48
Change from Baseline in Waist Circumference | Baseline, Week 32,Week 48
Percent Change from Baseline in Body Weight | Baseline, Week 48
Percentage of Participants who Achieve ≥5% Body Weight Reduction | Week 48
Percentage of Participants who Achieve ≥20% Body Weight Reduction | Week 32, Week 48
Change from Baseline in Neck Circumference | Baseline, Week 32, Week 48
Change from Baseline in Hip Circumference | Baseline, Week 32, Week 48
Change from Baseline in Body Weight | Baseline, Week 32, Week 48
Percent Change from Baseline in Body Weight | Baseline, Week 60
Change from Baseline in Body Mass Index (BMI) | Baseline, Week 32, Week 48
Percentage of Participants with BMI < 24 kg/m2 | Week 32, Week 48
Change from Baseline in Systolic Blood Pressure | Baseline, Week 32, Week 48
Change from Baseline in Diastolic Blood Pressure | Baseline, Week 32, Week 48
Change from Baseline in Triglyceride | Baseline, Week 32,Week 48
Change from Baseline in Total Cholesterol | Baseline, Week 32, Week 48
Change from Baseline in Low-density Lipoprotein Cholesterol | Baseline, Week 32, Week 48
Change from Baseline in High-density Lipoprotein Cholesterol | Baseline, Week 32, Week 48
Change from Baseline in Serum Uric Acid | Baseline, Week 32, Week 48
Change from Baseline in Alanine Aminotransferase | Baseline, Week 32, Week 48
Change from Baseline in Aspartate Aminotransferase | Baseline, Week 32, Week 48
Change from Baseline in Glycated Hemoglobin A1c (HbA1c) | Baseline, Week 32, Week 48
Change from Baseline in Fasting Plasma Glucose | Baseline, Week 32, Week 48
Change from Baseline in Fasting Insulin | Baseline, Week 32, Week 48
Change from Baseline in Fasting C-peptide | Baseline, Week 32, Week 48
Change from Baseline in Homeostatic Model Assessment of Insulin Resistance-Insulin Resistance Index (HOMA2-IR) | Baseline, Week 32, Week 48
Change from Baseline in IWQoL-Lite-CT Questionnaire Scores | Baseline, Week 32, Week 48
Change from Baseline in SF-36v2 Questionnaire Scores | Baseline, Week 32, Week 48

CONTACTS AND LOCATIONS:
Locations (23):
- China (23):
  - Xuancheng People's Hospital, Xuancheng, Anhui
  - People's Hospital of Peking University, Beijing, Beijing Municipality
  - Luoyang Third People's Hospital, Luoyang, He'nan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, He'nan
  - The First Affiliated Hospital of Nanyang Medical University, Nanyang, He'nan
  - The Third Affiliated Hospital of Xinxiang Medical University, Xinxiang, He'nan
  - Hebei Petro China Central Hospital, Langfang, Hebei
  - The First People's Hospital Of Kunshan, Kunshan, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Affiliated Hospital Of Nantong University, Nantong, Jiangsu
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - Shenyang Fifth People's Hospital, Shenyang, Liaoning
  - Jinan Central Hospital, Ji'nan, Shandong
  - Shandong Provincial Third Hospital, Ji'nan, Shandong
  - Qilu Hospital Of Shandong University (Qingdao), Qingdao, Shandong
  - Tai'an Central Hospital, Tai’an, Shandong
  - Zibo Municipal Hospital, Zibo, Shandong
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Yan'an University Xianyang Hospital, Xianyang, Shanxi
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - Lishui Central Hospital, Lishui, Zhejiang

REFERENCES:
- [Derived] Ji L, Jiang H, Bi Y, Li H, Tian J, Liu D, Zhao Y, Qiu W, Huang C, Chen L, Zhong S, Han J, Zhang Y, Lian Q, Yang P, Lv L, Gu J, Liu Z, Deng H, Wang Y, Li L, Pei L, Qian L; GLORY-1 Investigators. Once-Weekly Mazdutide in Chinese Adults with Obesity or Overweight. N Engl J Med. 2025 Jun 12;392(22):2215-2225. doi: 10.1056/NEJMoa2411528. Epub 2025 May 25. PMID 40421736